CLINICAL TRIAL: NCT06540261
Title: An Open-label, Uncontrolled Study of ONO-7913, ONO-4538 and the Standard of Care FOLFOX in Combination With Bevacizumab or Cetuximab as First-line Treatment in Patients With Unresectable Advanced or Recurrent Colorectal Cancer
Brief Title: The Study of ONO-7913, ONO-4538 and the Standard of Care as First-line Treatment in Patients Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONO-7913-04
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Unresectable Colorectal Cancer
MeSH Terms: interventions — magrolimab; Nivolumab; Fluorouracil; Oxaliplatin; Leucovorin; Bevacizumab; Cetuximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-7913＋ONO-4538＋FOLFOX＋Bev (Experimental)
  Interventions: Drug: ONO-7913; Drug: ONO-4538; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Bevacizumab
- ONO-7913＋ONO-4538＋FOLFOX＋Cet (Experimental)
  Interventions: Drug: ONO-7913; Drug: ONO-4538; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Cetuximab

INTERVENTIONS:
Drug: ONO-7913 — Specified dose on specified days
  Other Names: Magrolimab
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
Drug: Fluorouracil — Specified dose on specified days
Drug: Oxaliplatin — Specified dose on specified days
Drug: Levofolinate — Specified dose on specified days
Drug: Bevacizumab — Specified dose on specified days
  Arms: ONO-7913＋ONO-4538＋FOLFOX＋Bev
Drug: Cetuximab — Specified dose on specified days
  Arms: ONO-7913＋ONO-4538＋FOLFOX＋Cet

SUMMARY:
To confirm the tolerability and safety of combined administration of ONO-7913, ONO-4538 and the standard of care FOLFOX in combination with bevacizumab or cetuximab as first-line treatment in patients with unresectable advanced or recurrent colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable advanced or recurrent colorectal cancer
2. Life expectancy of at least 3 months
3. Patients with ECOG performance status 0 or 1

Exclusion Criteria:

1. Patients with severe complication
2. Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | 28 days
Adverse event (AE) | Up to 30 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics（Plasma concentration of ONO-7913） | Through study completion, an average of 1 year.
Pharmacokinetics（Plasma concentration of ONO-4538） | Through study completion, an average of 1 year.
Objective Response Rate (ORR) | Through study completion, an average of 1 year.
Disease Control Rate (DCR) | Through study completion, an average of 1 year.
Overall Survival (OS) | Through study completion, an average of 3 years.
Progression-Free Survival (PFS) | Through study completion, an average of 1 years.
Duration of Response (DOR) | Through study completion, an average of 1 years.
Time to Response (TTR) | Through study completion, an average of 1 years.
Best Overall Response (BOR) | Through study completion, an average of 1 years.
Percent change in the sum diameters of the target lesions | Through study completion, an average of 1 years.
Maximum percent change in the sum diameters of the target lesions | Through study completion, an average of 1 years.
Early Tumor shrinkage（ETS） | Up to 8 weeks
Change From Baseline in Tumour Biomarkers (CEA and CA19-9) | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (17):
- Japan (17):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Cancer Center, Shinden, Saitama
  - Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - National Cancer Center Hospital, Chūōku, Toyko
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: No